CLINICAL TRIAL: NCT05748106
Title: Comparison of a Novel Ultrasound System Versus Standard Imaging Modalities in the Context of Interventional Radiologic Procedures
Brief Title: Comparison of a Novel Ultrasound System Versus Standard Imaging Modalities
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: MAUI Imaging, Inc. (Industry)
Collaborators: Texas Health Resources (Other)
Responsible Party: Sponsor
Other Study IDs: 20203900a
Record Dates: First submitted 2023-02-07; First posted 2023-02-28 (Actual); Last update posted 2023-03-01 (Actual); Status verified 2023-02

CONDITIONS: Image-Guided Biopsies and/or Ablations
Keywords: Ultrasound Imaging; Interventional Radiology; Image-guided biopsy; Image-guided tumor ablation; Image-guided procedures

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: Ultrasound-based imaging — Ultrasound-based imaging
  Other Names: K3900

SUMMARY:
This is an observational study comparing a novel ultrasound-based imaging system (MAUI K3900) to standard-of-care (SoC) imaging systems used to guide and/or manage interventional radiologic procedures such as solid organ biopsies or lesion ablations.

DETAILED DESCRIPTION:
The purpose of this study is to obtain images using the MAUI Imaging Inc.'s K3900 Ultrasound System and compare them to images captured with FDA cleared imaging devices including traditional ultrasound, CT, MRI and Xray, and to study device safety. The information obtained in this study will inform MAUI Imaging as to what specific follow-on studies will be done in support of appropriate FDA clearances and/or claims. No diagnostic or patient management decisions will be made using the MAUI K3900 Ultrasound System in this study.

ELIGIBILITY:
Inclusion Criteria:

* Undergoing standard / routine interventional radiologic procedure

Exclusion Criteria:

* Unwilling or unable to provide informed consent

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Any patient undergoing a standard / routine interventional radiologic procedure
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2023-02-15 (Actual); Primary Completion 2023-05-30 (Estimated); Study Completion 2023-06-30 (Estimated)

PRIMARY OUTCOMES:
Usefulness relative to standard imaging for image-guided solid organ biopsies and/or ablations | Up to 26 weeks
  How does imaging with the K3900 compare with imaging currently used to guide solid organ biopsies or ablations, usually standard ultrasound, fluoroscopy, and/or CT?

CONTACTS AND LOCATIONS:
Overall Officials: John C Cheronis, MD/PhD, Study Director — MAUI Imaging, Inc.
Locations (1):
- Texas Health Presbyterian Hospital, Dallas, Texas, United States

IPD SHARING:
Plan to Share IPD: No